CLINICAL TRIAL: NCT02309866
Title: Identifying Genes and Mutations Underlying Retinitis Pigmentosa and Allied Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 83-13
Record Dates: First submitted 2014-11-24; First posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-11

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — genomic DNA

GROUPS / COHORTS (1):
- Genetic Testing: All participants determined eligible for the study will be placed into genetic testing arm.
  Interventions: Genetic: Genetic testing

INTERVENTIONS:
Genetic: Genetic testing — Genetic testing for mutations in known and novel genes underlying RP and allied diseases

SUMMARY:
Retinitis Pigmentosa (RP) is the most common form of hereditary retinal degeneration, with a worldwide prevalence of 1:3500. It is one of the most genetically heterogenous conditions in humans, with over 100 causative genes and loci reported to date. However, in approximately 40% of patients the underlying genetic causes are yet to be found.

The current study aims to identify causative RP genes and mutations in Israeli families of various ethnic backgrounds. Identification of such genes will contribute significantly to disease prevention (by identification of high risk families and appropriate genetic counseling) and to the investigators understanding of retinal structure and function and of the etiology of RP.

DETAILED DESCRIPTION:
Background: Retinitis Pigmentosa (RP) is a clinically and genetically heterogeneous disease, which causes visual loss due to the premature death of retinal photoreceptors. Over 100 genes and loci have been implicated in RP. However, the contribution of each of these genes to the overall prevalence of RP is relatively small, and many of them are yet to be found. These unidentified genes are likely to be very rare. The vast majority of studies on the genetics of RP have been performed on the American and European populations. Based on the investigators experience, the genetic makeup of the Israeli population is unique, and many of the genetic alterations identified in Israeli patients are novel.

Working hypothesis and aims: the investigators working hypothesis is that the Israeli population is unique in terms of the identity and relative contribution of RP genes. Therefore, the investigators aim is to perform a comprehensive genetic analysis of affected Israeli individuals of various ethnic backgrounds, in order to identify novel RP mutations and genes.

Methods: RP patients and family members will be continuously recruited to the study through the Ophthalmology Department at Hillel Yaffe Medical Center, Hadera, Israel. The relatively high proportion of founder mutations in the Israeli population allows us to perform a quick and efficient mutation screening and identify the cause of disease in a large number of newly recruited families. Patients who are negative for all relevant mutations will be studied using whole exome sequencing. Bioinformatic analysis will be used to identify possible pathogenic variants. Following verification, the investigators will check their co-segregation with the disease in the entire family, and their frequency in the relevant population.

Expected results: The immediate expected outcomes include an epidemiological overview of RP distribution and etiology in the Israeli population, and identification of novel causative genes and mechanisms. These genes are expected to play a crucial role in retinal development and function, and hence their identification and characterization will contribute significantly to the investigators understanding of retinal structure and function and of the etiology of RP. The main expected long-term outcome is reduction in the frequency of RP in Israel. This will be achieved by a combination of prevention (by genetic screening and counseling among high-risk populations), and treatment (by identification of patient groups with shared genetic diagnoses, who can be recruited to clinical trials for evaluation of various treatment strategies).

ELIGIBILITY:
Inclusion Criteria:

* Patients with RP in which the genetic cause has not been identified yet and their healthy family members

Exclusion Criteria:

* Patients with RP in which the genetic cause has already been identified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be composed of Israeli individuals who have been clinically diagnosed with RP but do not have a confirmed diagnosis by genetic testing.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Percent of patients in whom common founder mutations in known RP-related gene are found | 4 years
Percent of patients in whom mutations in novel RP-related genes are found | 4 years